CLINICAL TRIAL: NCT05009095
Title: The Listening Program With Bone Conduction Headphones Changes Hypersensitivity to Sound and Behavioral Responses Associated With Flight/Fight Responses of Children With Autism Spectrum Disorder Therefore Increasing Adaptive Life Skills
Brief Title: The Listening Program® With Bone Conduction Headphones Changes Hypersensitivity to Sound and Behavioral Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Health (Other)
Responsible Party: Principal Investigator, Suzanne Vercontaire, Occupational Therapist III, Children's Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-1698
Record Dates: First submitted 2021-08-03; First posted 2021-08-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; The Listening Program® with bone conduction headphones; Hypersensitivity to sound and behavioral responses
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The study will use a nonconcurrent AB multiple baseline design, with A representing the baseline phase and B representing the intervention phase with a postintervention non-treatment phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- The Listening Program® with bone conduction headphones (Experimental): The Listening Program ® Spectrum music requires a person listen to psycho-acoustically modified classical music online using specialized "Waves" ™ headphones. The headphones transmit sound through bone conduction which provides another mode of perceiving sound (https://advancedbrain.com). The Listening Program ® can be carried out in the home environment with either the base schedule, two fifteen minute sessions at least 30 minutes apart, or a condensed schedule for 30 minutes.
  Bone conduction allows the listening experience to go deeper into the vestibular system which is purported to reduce stress, help regulate the "fight or flight" response, and allow the listener to achieve a state of calm and relaxed alertness. This theory is based on the function of the vagus nerve, the 10th cranial nerve, which has branches that extend to the eardrum. Stimulation of the vagus nerve stimulates the parasympathetic nervous system (Allen, 2008).
  Interventions: Device: The Listening Program® with bone conduction headphones

INTERVENTIONS:
Device: The Listening Program® with bone conduction headphones — The Listening Program method of Music-Based Auditory Stimulation is enhanced with the addition of bone conduction technology with the ABT Bone Conduction System. Bone Conduction combines the experience of listening to music through modified headphones adding subtle, synchronized acoustic vibration of the skin and skeletal system, engaging the whole body and brain in the listening process. This multi-sensory approach accelerates and expands the benefits of The Listening Program.

SUMMARY:
There are limited approaches to specifically address auditory sensory over- and under-responsivity (SOR) in children with Autism Spectrum Disorder (ASD). Exposure therapy (or systematic desensitization) may be a treatment option; researchers are investigating this approach. Many children receive sensory integration therapy, but this approach does not specifically target auditory SOR. Some families are advised to have their children avoid noxious stimuli or use compensatory techniques such as wearing headphones or ear plugs. While preliminary research suggests that use of noise attenuating headphones may reduce sympathetic activation for children with ASD and auditory SOR, this approach does not seek to change or alter the underlying cause of sympathetic activation (Pfeiffer et al., 2019).

Sound-based interventions are promising options to treat hyperacusis and subsequent auditory SOR in children with ASD. The objective of this study is to investigate changes in adaptive life skills and behavioral responses in children with ASD using Advanced Brain Technology's The Listening Program ® Spectrum music utilizing Waves ™ (bone conduction) headphones.

Our study will investigate the effects of a sound-based intervention developed in 2012 to specifically address the needs of children with ASD and children with hyperacusis and/or auditory SOR - The Listening Program® Spectrum music utilizing Waves™ (bone conduction) headphones by Advanced Brain Technologies. This program emphasizes low frequency music over an extended period of time; the duration recommended by Advanced Brain Technologies is 40 weeks.

DETAILED DESCRIPTION:
Children with a diagnosis of ASD with auditory SOR to sound, ages 5 to 10 years, will be the primary patient population. The study will use a nonconcurrent AB multiple baseline design, with A representing the baseline phase and B representing the intervention phase with a postintervention non-treatment phase. At baseline (A), demographic information will be collected and the following outcome measures will be completed: the Pediatric Evaluation of Disability Inventory Computer Adaptive Test with ASD Scales (PEDI CAT- ASD), Sensory Processing Measure (SPM) home form, the Adaptive Behavioral Assessment System 3rd Edition ABAS-3 and Autism Treatment Evaluation Checklist (ATEC). During the intervention (B) phase, parents of participants in the treatment group will be educated by the investigators on use of The Listening Program at home, and then participants in this group will receive treatment at home utilizing The Listening Program for 40 weeks. Testing, using the same 4 outcome measures, will be completed at the 41st week after use, and then again after 3 months of no treatment. Between testing sessions, caregivers and investigators will set up three phone or hospital-approved virtual platform meetings at approximately 10 week intervals to check in and answer questions.

ELIGIBILITY:
Inclusion Criteria:

1. Children will be eligible to participate in this study if they are:

1. Between the ages of 5 and 10 years old
2. Diagnosis of autism spectrum disorder
3. Auditory SOR defined by "Some Problems or Definite Dysfunction" on the Hearing section on the Sensory Processing Measure Home Form.
4. Caregiver must be available to supervise listening sessions at home
5. English Speaking

Exclusion Criteria:

1. Children will be excluded from the study if they are:

a. Diagnosed with seizure disorder b. Hearing impairments c. Cerebral palsy d. Fragile X syndrome or genetic disease e. Previous use of a listening base system f. Non-English speakers

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Adaptive Behavior Assessment System, Third Edition (ABAS-3) Score at 41 Weeks (Immediately Post-Treatment) | To be administered at baseline, 1-week following a 40-week use of the listening program.
  The third edition of this highly regarded assessment gives a complete picture of adaptive skills across the life span. Per the test manual, the ABAS-3 has good test-retest reliability (r .72 - .84 across all areas/domains). The ABAS-3 is easy to administer and score. It is particularly useful for evaluating those with developmental delays, autism spectrum disorder, intellectual disability, learning disabilities, neuropsychological disorders, and sensory or physical impairments (Harrison & Oakland, 2015). The ABAS-3 covers individuals from birth to 89 years of age (www.wpspublish.com/)

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory Computer Adaptive Test with ASD Scales (PEDI-CAT (ASD)) | To be administered at baseline, 1-week following a 40-week use of the listening program, and 3-months following treatment
  The PEDI-CAT (ASD) is a module of the PEDI-CAT that has been validated for the population of children and adolescents with ASD. The PEDI-CAT (ASD) includes directions to help parents select an appropriate rating given the unique characteristics of children with autism. This module also includes new or revised items in the Daily Activities, Social/Cognitive, and Responsibility domains.
  The PEDI-CAT does not require any special environment, materials or activities for administration. The PEDI-CAT can be completed directly by the child's caregiver(s) or by the child's therapist/clinician. The assessment focuses on typical performance at the present time.
  The PEDI-CAT can be used on multiple occasions for the same child (e.g. initial, interim, discharge and follow-up) and there is no minimum time that must pass between assessments.

OTHER OUTCOMES:
Sensory Processing Measure™ (SPM™) | To be administered at baseline, 1-week following a 40-week use of the listening program, and 3-months following treatment
  The Sensory Processing Measure (SPM) is a norm-referenced assessment of sensory integration/sensory processing that gathers information about a child's behavior, coordination, and participation at home, in the community, and/or at school. For the purposes of the study the Home Form will be utilized. Per test manual, the SPM has good test-retest reliability (r ≥.94 on all scales). Separate scores are provided for social participation, five sensory systems, and motor planning in the home. Additional scores may be obtained for six different school settings, including art class, music class, physical education class, the playground, the cafeteria, and the school bus. Sensory Processing Measure (SPM) can be used with 5- to 12-year-old children, including 5-year-olds who have already started kindergarten (Parkham, Kuhaneck, Henry & Glennon, 2007)
Autism Treatment Evaluation Checklist (ATEC) | To be administered at baseline, 1-week following a 40-week use of the listening program, and 3-months following treatment
  The ATEC is a 77-item assessment tool developed at the Autism Research Institute. It was developed to provide a free, easily accessible, and valid tool to measure changes in ASD symptoms over time. The ATEC can be completed by parents, teachers, or others who see the individual's behavior on a regular basis. The ATEC consists of four subtest scales: Speech/Language/Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical Behavior. The four subscale scores are used to calculate a total score (77 items - score range 0 to 180). A lower score indicates less severe symptoms of ASD and a higher score correlates with more severe symptoms of ASD. Baseline scores can be compared with post-intervention scores to assist with determining intervention efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Vercontaire, Principal Investigator — Children's Health
Locations (1):
- Childrens's Health Specialty Center Richardson, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kramer JM, Liljenquist K, Coster WJ. Validity, reliability, and usability of the Pediatric Evaluation of Disability Inventory-Computer Adaptive Test for autism spectrum disorders. Dev Med Child Neurol. 2016 Mar;58(3):255-61. doi: 10.1111/dmcn.12837. Epub 2015 Jun 22. PMID 26104112